CLINICAL TRIAL: NCT00751387
Title: Australian Descriptive Epidemiology Study of Severity of Rheumatoid Arthritis (RA), Psoriatic Arthritis (PsA) and Ankylosing Spondylitis (AS) and Exposure to Biological Disease Modifying Anti-rheumatic Drugs (bDMARDs)
Brief Title: Study Evaluating Epidemiology of Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis in Australia
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0881X1-4519; B1801088
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Ankylosing Spondylitis; Psoriatic Arthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The study is a cross sectional, epidemiology study of disease severity for rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis in four geographic regions in Australia (Illawarra, Sutherland, Hunter Urban and Hunter Rural).

ELIGIBILITY:
Inclusion criteria include:

Adult patients with a diagnosis of rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis who have visited a primary care centre within one of the specified catchment areas for their condition within the last 24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Proportion of rheumatoid arthritis/psoriatic arthritis/ankylosing spondylitis patients in defined disease severity categories | Single visit

SECONDARY OUTCOMES:
Proportion of patients exposed to biological disease modifying antirheumatic drugs | Single visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- Australia (4):
  - Georgetown
  - Miranda
  - Newcastle
  - Wollongong